CLINICAL TRIAL: NCT00910845
Title: Study of Botulinum Toxin Type A for the Treatment of Patients With Idiopathic Overactive Bladder With Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-095
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- onabotulinumtoxinA (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 100 U injected into the detrusor at Day 1, followed by a repeat injection of onabotulinumtoxinA 100 U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA
- placebo/onabotulinumtoxinA (Other): Placebo (normal saline) injected into the detrusor at Day 1, followed by an injection of onabotulinumtoxinA (botulinum toxin Type A) 100 U after a minimum of 12 weeks (if applicable).
  Interventions: Biological: onabotulinumtoxinA; Drug: normal saline

INTERVENTIONS:
Biological: onabotulinumtoxinA — OnabotulinumtoxinA (botulinum toxin Type A) 100 U injected into the detrusor at Day 1, followed by a repeat injection of onabotulinumtoxinA 100 U after a minimum of 12 weeks (if applicable). Or, if placebo is administered at Day 1, onabotulinumtoxinA 100 U injected after a minimum of 12 weeks (if applicable).
  Other Names: BOTOX®; botulinum toxin Type A
Drug: normal saline — Normal saline (placebo) injected into the detrusor at Day 1.
  Arms: placebo/onabotulinumtoxinA

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of botulinum toxin type A (onabotulinumtoxinA) in treating patients with idiopathic overactive bladder with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of OAB (frequency/urgency) with urinary incontinence for at least 6 months
* Inadequate response or limiting side effects with anticholinergics for the treatment of OAB

Exclusion Criteria:

* Overactive Bladder caused by neurological condition
* Patient has predominance of stress incontinence
* History or evidence of pelvic or urological abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Newport Beach, California, United States
- Victoria, British Columbia, Canada

REFERENCES:
- [Derived] McCammon K, Gousse A, Kohan A, Glazier D, Gruenenfelder J, Bai Z, Patel A, Hale D. Early and Consistent Improvements in Urinary Symptoms and Quality of Life With OnabotulinumtoxinA in Patients With Overactive Bladder and Urinary Incontinence: Results From a Randomized, Placebo-controlled, Phase IV Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Jul 1;27(7):450-456. doi: 10.1097/SPV.0000000000000914. PMID 32665528
- [Derived] Castejon N, Khalaf K, Ni Q, Cuervo J, Patrick DL. Psychometric properties of the incontinence utility index among patients with idiopathic overactive bladder: data from two multicenter, double-blind, randomized, Phase 3, placebo-controlled clinical trials. Health Qual Life Outcomes. 2015 Aug 1;13:116. doi: 10.1186/s12955-015-0306-5. PMID 26231052
- [Derived] Sievert KD, Chapple C, Herschorn S, Joshi M, Zhou J, Nardo C, Nitti VW. OnabotulinumtoxinA 100U provides significant improvements in overactive bladder symptoms in patients with urinary incontinence regardless of the number of anticholinergic therapies used or reason for inadequate management of overactive bladder. Int J Clin Pract. 2014 Oct;68(10):1246-56. doi: 10.1111/ijcp.12443. Epub 2014 Apr 22. PMID 24754838

RESULTS

PARTICIPANT FLOW:
Period: Treatment Cycle 1
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Started | 280 | 277
Completed | 249 | 243
Not Completed | 31 | 34
Period: Treatment Cycle 2
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Started | 141 (Not all participants who completed Treatment Cycle 1 went onto Treatment Cycle 2) | 212 (Not all participants who completed Treatment Cycle 1 went onto Treatment Cycle 2)
Completed | 136 | 203
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA | Total
Number analyzed (Participants) | 280 | 277 | 557
Age, Customized [Number; unit: Participants]
  < 40 years | 9 | 17 | 26
  Between 40 and 64 years | 150 | 143 | 293
  Between 65 and 74 years | 75 | 73 | 148
  ≥ 75 years | 46 | 44 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 245 | 497
  Male | 28 | 32 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Number of Daily Episodes of Urinary Incontinence
Description: A urinary incontinence episode is defined as an incident of involuntary loss of urine as recorded in a patient bladder diary during the 3 days before the Baseline and Week 12 study visits. A negative number change from baseline indicates a reduction in incontinence episodes (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: Incontinence episodes
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 280 | 277
Incontinence episodes
  Baseline | 5.47 (3.621) | 5.09 (3.204)
  Change from Baseline at Week 12 | -2.65 (3.333) | -0.87 (2.833)

2. Secondary Outcome: Change From Baseline in Number of Daily Micturition Episodes
Description: The number of micturition episodes (the number of times a patient urinates into the toilet) was recorded by the patient in a bladder diary during 3 consecutive days in the week prior to the Baseline and prior to the Week 12 study visit. A negative number change from baseline indicates a reduction in micturition episodes (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: micturition episodes
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 280 | 277
micturition episodes
  Baseline | 11.98 (4.259) | 11.20 (3.070)
  Change from Baseline at Week 12 | -2.15 (2.933) | -0.91 (2.577)

3. Secondary Outcome: Change From Baseline in Volume Voided Per Micturition
Description: The total volume voided was measured over one 24-hour period in the week prior to the Baseline and Week 12 study visit and recorded by the patient in the bladder diary. This was used to calculate volume voided per micturition. A positive number change from baseline indicates an increase in volume voided per micturition (improvement).
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all randomized patients.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Number analyzed (Participants) | 280 | 277
milliliters
  Baseline | 156.4 (63.21) | 161.1 (68.65)
  Change from Baseline at Week 12 | 41.1 (87.58) | 9.7 (59.02)

ADVERSE EVENTS:
Description: The safety population was used to calculate the number of participants at risk for Serious Adverse Events (SAEs) and Adverse Events (AEs) and is the total number of patients who were treated. S(AE)s are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | onabotulinumtoxinA | Placebo/onabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 18/278 | 16/272
Other Adverse Events (participants affected / at risk) | 155/278 | 79/272
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA (N=278) | Placebo/onabotulinumtoxinA (N=272)
Coronary artery disease (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Foramen magnum stenosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Obesity (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 2 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | onabotulinumtoxinA (N=278) | Placebo/onabotulinumtoxinA (N=272)
Urinary tract infection (Infections and infestations) | 68 | 25
Bacteriuria (Infections and infestations) | 23 | 10
Dysuria (Renal and urinary disorders) | 40 | 27
Urinary retention (Renal and urinary disorders) | 16 | 1
Haematuria (Renal and urinary disorders) | 8 | 16 — Event not treatment related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.